CLINICAL TRIAL: NCT02548702
Title: Effect of a Community-based Sport Programme on Disease Symptoms and Quality of Life in Men and Women With Type 2 Diabetes
Brief Title: Community-based Sport Programme and Type 2 Diabetes
Acronym: Fit4Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: Community Sport Trust (Unknown); Sport Nottinghamshire (Unknown); Sport England (Other); Nottingham City Clinical Commissioning Group (Other); NHS North and East Nottinghamshire Clinical Commissioning Group (Other); NHS Lincolnshire West Clinical Commissioning Group (Other); NHS Rushcliffe Clinical Commissioning Group (Other); Nottingham City Council (Unknown); Nottinghamshire County Council (Unknown)
Responsible Party: Principal Investigator, Prof. Mary Nevill, Professor and Head of Department of Sport Science, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTU2290
Record Dates: First submitted 2015-09-03; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes
Keywords: Sport; type 2 diabetes; community intervention programme; Fit4life; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community-based sport (Experimental): Patients with type 2 diabetes will receive motivational counselling and will be allocated to a low intensity community-based sporting activity (Fit4Life programme) depending on their interests and perceived barriers to taking part.
  Interventions: Behavioral: Fit4Life
- Control (No Intervention): One in 10 participants will be allocated to a control group who do not receive the intervention

INTERVENTIONS:
Behavioral: Fit4Life — Fit4Life is a programme whereby patients with type 2 diabetes are counselled and then allocated to a community-based sport programme based on their interests and perceived barriers to participation
  Arms: Community-based sport

SUMMARY:
The Fit4Life intervention aims to engage inactive patients with type 2 diabetes in a community-based sport intervention, with the aim being that all participants complete 1 x 30 min session of physical activity/exercise per week across the 12 months they are involved in the intervention (total study duration 3 years).

The aim of the Fit4Life intervention is to slow the progression of disease symptoms and to improve quality of life in those diagnosed with type 2 diabetes. The aim of this research study is thus to evaluate the effectiveness of the intervention in achieving these aims. The hypothesis is that involvement in the Fit4Life programme will increase physical activity, reduce type 2 diabetes disease symptoms and enhance self-reported quality of life in male and female patients aged 35-64.

DETAILED DESCRIPTION:
Overview The evaluation will also assess the effect of the community-based sport intervention (1 x 30 min session per week) on physical activity levels and cognitive function in type 2 diabetes patients. Physical activity is known to assist in the management of type 2 diabetes, thus the effect of the intervention on physical activity levels is of interest. In addition, type 2 diabetes has been shown to detrimentally affect cognitive function. Therefore, the evaluation will also assess the effect of the community-based sport intervention on cognitive function in the type 2 diabetes patients.

This project will engage inactive patients diagnosed with type 2 Diabetes in regular sport and physical activity. The aim of the project is to use community based sport and physical activity to enhance health and wellbeing and to facilitate the effective management of type 2 diabetes. Working in Nottingham City with 60 GP Practices and their Diabetes Specific Nurses, and in the 3 south area CCGs with up to 60 GP Practices, patients' sporting interests and motivations will be identified and matched with appropriate, local, community-based sport and exercise opportunities delivered by specially trained instructors and coaches. The aim of the study (total duration 3 years) is to engage 4032 people in 1 x 30 minutes of sport/exercise per week, for 12 months.

Primary research question(s)/evaluation aim(s):

Change from baseline in number of participants reporting one or more sessions of sport per week measured by the UK Single Item Questionnaire.

Secondary research question(s)/evaluation aim(s):

Change from baseline in body mass (kg); Change from baseline in hip circumference (cm) Change from baseline in waist circumference (cm) Change from baseline in quality of life as measured by the Quality of Life Survey (QOLS)(sum of 16 item, 7 point likert scale); Change from baseline in control of blood glucose concentration as measured by self-report survey(subjective rating, 'better', 'the same', 'worse'); Change from baseline in control of blood glucose concentration as measured by HPA1c concentration (mmol/mol)

Objectives To use community based sport and physical activity to engage 4032 inactive patients, diagnosed with type 2 diabetes, in 1 x 30 minutes of sport / exercise per week, over 3 years. In so doing, to enhance the health and wellbeing of the patients and to help facilitate the effective management of their type 2 diabetes.

Design A questionnaire will be distributed to 4032 patients (over the 3 year duration of the project) at baseline, 3, 6 and 12 months. The questionnaire will ask questions about sports participation, physical activity undertaken and sedentary behaviour, which will allow examination of whether the Fit4life project has increased the quantity of sport and physical activity undertaken by inactive patients, diagnosed with type 2 diabetes. The questionnaire will also contain questions investigating the quality of life of patients, perception of effort and the type and quantity of medication used by patients during their involvement in the Fit4 life project; this will allow examination of whether the Fit4life project has enhanced the health and wellbeing of inactive patients, diagnosed with type 2 diabetes.

In addition, as per Sport England requirements, data will be collected on: The number of people engaged with the project (target and outcome measure); the number of inactive people engaged in the project; the number of inactive people moved into 1 x 30 minutes of sport; the number of people still engaged in the sport at 3, 6 and 12 months.

In a small sub-sample of patients involved in the project (n=50-100) some direct assessments of physical activity, health status and physiological function will be made. These assessments may include measurement of: physical activity via accelerometers / pedometers; waist and hip circumference; fasting blood glucose, HPA1c and c-peptide concentrations; responses to treadmill walking.

In order to provide rich, explanatory data, to provide information about project processes, and how the project worked and was received, focus groups / telephone interviews will be conducted with patients (n=30-40 per year), practitioners and key stakeholders.

The survey will include questions on:

* The number of people engaged with the project
* The number of inactive people engaged in the project
* The number of inactive people moved into 1 x 30 minutes of sport
* The number of people still engaged in the sport at 3 months
* The number of people still engaged in the sport at 6 months
* The number of people still engaged in the sport at 12 months
* Socio-economic status via post code and income
* Demographic characteristics e.g. sex, ethnicity, religion and disability
* Perception of effort via a Borg scale
* Quality of life
* Diabetes medication use
* Diabetes symptoms
* Enjoyment of sporting sessions
* Quality of sporting sessions, leader, venue, intensity and duration

Measured directly in all participants by the project team:

* Waist and hip circumference
* Height and body mass

Measured directly by the investigators in a sub-sample of 50-100:

* physical activity via accelerometers / pedometers
* waist and hip circumference
* height and body mass
* fasting blood glucose
* HPA1c and c-peptide concentrations
* responses to treadmill walking

Focus groups and telephone semi-structured interviews in a sub-sample of 40-50 participants (accepted qualitative methods)

* Process evaluation
* Perceptions of health and fitness as a result of project participation

Approximately four thousand patients will be recruited to the project and randomly allocated to an experimental group (9/10 patients recruited at each time point) and a control group (1/10 patients recruited at each time point). The experimental group will complete the questionnaire at 0, 3, 6 and 12 months of involvement with the Fit4Life project. The control group will complete the questionnaire at 0 and 3 months. Due to the need to provide a service to all participants and to solicit the co-operation of GPs involved with the project the control participants will then join the sporting activities offered to all other participants, but will take no further part in the evaluation. As control participants will be recruited throughout the project, statistically their data will be combined to form a rolling control for the full period of the intervention and the analysis will be a mixed longitudinal design undertaken by a consultant statistician (Prof. Alan Nevill).

Patients will be recruited from approximately 240 GP practices in the Nottingham City and South Nottinghamshire area. GPs will provide patients with the project information (including a telephone and email contact number) and patients will contact the project team themselves. Patients can also self-refer from road shows and other events but will be asked to obtain a note from their GP expressing their suitability to take part in the project.

A process evaluation (how has the project worked for staff and patients) will be undertaken via focus groups and telephone interviews as described earlier.

Time-scale September/October 2015: NHS Ethics approval gained October 2015 onwards: patient recruitment to intervention and control groups on-going throughout the study October 2015: first patients recruited complete the baseline questionnaire and the intervention group have their motivational interview October 2015: intervention group start sporting activities December 2015: the earliest recruited control and intervention group patients complete the 3 month survey; the first controls join the sporting activities but take no further part in the evaluation February 2016: first focus groups with patients and interviews with leaders and staff take place March 2016: the earliest recruited intervention group patients complete the 6 month survey May 2016: further focus groups and interviews take place June 2016: the earliest recruited intervention group patients complete the 9 month survey September 2016: the earliest recruited intervention group patients complete the 12 month survey September 2016: end of year one report submitted to Sport England October 2016: dissemination of early findings September 2017: end of year two report submitted to Sport England October 2017: dissemination of interim findings September 2018: final report submitted to Sport England October 2018: dissemination of study findings

Analysis of results Survey data will be downloaded to SPSS (Statistical package for the Social Sciences) and the differences between the intervention and control group (accounting for sex and demographic characteristics) will be examined using an appropriate statistical methods such as multi-level modelling with a mixed longitudinal design.

Interview and focus group data will be transcribed, coded and analysed by interview themes and by themes (including unexpected outcomes) that emerge from the data set.

Laboratory data will be directly analysed using standard laboratory procedures such as the determination of oxygen uptake from expired air samples and the determination of blood glucose using an automated PENTRA analyser with purchased standards and controls.

All patients recruited to the Fit4life programme will have an initial assessment during which the baseline questionnaire will be completed. This assessment will take place at a GP clinic. Patients will start the study in groups of 10 to ease the logistical problems of follow-up measurements. Patients will have a further introduction to the study (verbal and written) in addition to the initial information received by telephone and in a written format on recruitment. Patients will sign an informed consent form and will complete the baseline questionnaire (with the opportunity to ask questions to project staff). In addition the intervention and the control group will have body mass, height, waist and hip circumference measured in private by project staff. Control participants will leave once the baseline questionnaire and anthropometric measurements have been completed and will return after 3 months to complete another questionnaire and to join the sporting activities (these participants will not be included in the intervention group for the evaluation). Patients will also have been asked to weigh themselves on home scales before they arrive. Project staff will then undertake the motivational interview with the intervention group participants and they will be allocated to a sporting activity.

Thus all participants recruited should complete the baseline survey. To enhance the completion of the 3 month and subsequent surveys, these will be administered at sporting venues where possible (and where facilities are available) by project staff who the patients have got to know. Where this is not possible patients will be invited back to the original clinic by project staff who they have got to know through the motivational interview. Surveys will be posted or emailed out to patients who are not caught by either of these methods. A limitation here is that participants will have to weigh themselves in their own homes, but we will have obtained a validation measure of their scales via the initial assessment meeting.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic
* inactive

Exclusion Criteria:

* taking part in regular sport or physical activity (more than 30 minutes on one day per week)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4032 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in number of participants reporting one or more sessions of sport per week measured by the UK Single Item Questionnaire | 3 years

SECONDARY OUTCOMES:
Change from baseline in body mass (kg) | 3 years
Change from baseline in hip circumference (cm) | 3 years
Change from baseline in waist circumference | 3 years
Change from baseline in quality of life as measured by the quality of life survey (QOLS)(sum of 16 item 7 point likert scale) | 3 years
Change from baseline in control of blood glucose concentration as measured by self-report survey (subjective rating, 'better', 'the same', 'worse' | 3 years
Change from baseline in control of blood glucose concentration as measured by HPA1c (mmol/mol) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Nevill, PhD, Principal Investigator — Nottingham Trent University
Locations (1):
- Nottingham Trent University, Nottingham, United Kingdom

REFERENCES:
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588